CLINICAL TRIAL: NCT02909465
Title: A Comparison of Midazolam or Haloperidol Premedication Versus Placebo for Reducing Ketamine Induced Agitation After Adult Procedural Sedation in the Emergency Department
Brief Title: Reducing Ketamine-Induced Agitation, by Midazolam or Haloperidol Premedication After Adult Procedural Sedation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Pooya Payandemehr, assistant professor of emergency medicine, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TehranUMS-ketamine
Record Dates: First submitted 2016-07-28; First posted 2016-09-21 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-03

CONDITIONS: Ketamine Induced Agitation
MeSH Terms: interventions — Midazolam; Haloperidol; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo (Placebo Comparator): To do procedural sedation and analgesia in this group, the patients will receive 2 intravenous injections of distilled water (one 2 ml and the other 0.05 cc/kg) 5 minutes before receiving a sedative dose of 1 mg/kg IV ketamine.
  Interventions: Drug: placebo; Drug: Ketamine
- midazolam (Experimental): To do procedural sedation and analgesia in this group, the patients will receive 2 intravenous injections. one will be 2 ml of distilled water and the other 0.05 mg/kg midazolam, 5 minutes before receiving a sedative dose of 1 mg/kg IV ketamine.
  Interventions: Drug: Midazolam; Drug: placebo; Drug: Ketamine
- haloperidol (Experimental): To do procedural sedation and analgesia in this group, the patients will receive 2 intravenous injections. One will be 0.05 cc/kg of distilled water and the other 5 mg of haloperidol (in 2 cc syringes), 5 minutes before receiving a sedative dose of 1 mg/kg IV ketamine.
  Interventions: Drug: Haloperidol; Drug: placebo; Drug: Ketamine

INTERVENTIONS:
Drug: Midazolam — Using Midazolam as a premedication for reducing ketamine-induced agitation
  Other Names: verdes
  Arms: midazolam
Drug: Haloperidol — Using Haloperidol as a premedication for reducing ketamine-induced agitation
  Other Names: haldol
  Arms: haloperidol
Drug: placebo — distilled water
Drug: Ketamine — Ketamine is routinely used for all procedural sedation in the patients.
  Other Names: ketalar

SUMMARY:
Ketamine is the cornerstone of procedural sedation in emergency department but ketamine induced agitation has limited its usage by many physicians. As a solution, some propose using midazolam or haloperidol before ketamine injection. In this randomized double blind clinical trial, patients who are eligible for sedation by ketamine are allocated in 3 groups. In first group, the patients will receive 0.05 mg/kg midazolam, in second group 5 mg of haloperidol and in 3rd group a placebo five minutes before receiving the sedative dose of ketamine (1 mg/kg). The patients are assessed for agitation during and after the procedure the clinician's satisfaction with sedation instrument is evaluated after the procedure.

DETAILED DESCRIPTION:
Ketamine is the cornerstone of procedural sedation in emergency department but ketamine induced agitation has limited its usage by many physicians. As a solution, some propose using midazolam or haloperidol before ketamine injection. In this randomized double blind clinical trial, patients who are eligible for sedation by ketamine are allocated in 3 groups. In first group, the patients will receive 0.05 mg/kg midazolam, in second group 5 mg of haloperidol and in 3rd group a placebo five minutes before receiving the sedative dose of ketamine (1 mg/kg). The patients are assessed for agitation during and after the procedure the clinician's satisfaction with sedation instrument is evaluated after the procedure. The investigator will fill standard questionnaires for agitation assessment (Richmond Agitation-Sedation Scale and Pittsburgh Agitation Scale).

ELIGIBILITY:
Inclusion Criteria:

* adult patient older than 18, who need to sedate in Emergency Department

Exclusion Criteria:

* age younger than 18 years,
* patients with significant cardiovascular disease,congestive heart failure (CHF)
* central nervous system lesions or injuries, increased intracranial pressure (ICP)
* ocular pathology, increased intraocular pressure (IOP)
* thyroid disease,
* acute pulmonary infections,
* conditions requiring stimulation of the posterior pharynx,
* had ingested solid food in the previous 4 hours or clear liquids in the previous 2 hours.
* Acute intermittent porphyria
* Alcoholism
* Hepatic Impairment
* Myasthenia gravis
* Respiratory depression
* allergy to haloperidol as established by direct questioning of family members and available medical history,
* moderate to severe dementia as documented by medical history,
* Parkinson's disease,
* corrected QTc interval (QTc) greater than 500 ms,
* usage of drugs prolonging QT-interval,
* history of torsades de pointes,
* history of neuroleptic malignant syndrome,
* family history of dystonic reactions to drugs,
* epilepsy or history of seizures
* chronic psychiatric disease,
* intoxication
* bone marrow suppression
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2016-07; Primary Completion 2017-04 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
agitation | starts at the time of Ketamine injection through recovery period(maximum of 2 hours)
  assessed by Pittsburgh Agitation Scale(scoring 0 to 16).
  Pittsburgh Agitation Scale(scoring 0 to 16) is a valid and reliable instrument to assess agitation severity of inpatients.
level of sedation | 5 minutes after Ketamine injection
  assessed by Richmond Agitation-Sedation Scale(scoring -5 to +4).
  Richmond Agitation-Sedation Scale(scoring -5 to +4) is a valid and reliable instrument to assess level of sedation and agitated behavior during sedation.
level of sedation | 15 minutes after Ketamine injection
  assessed by Richmond Agitation-Sedation Scale(scoring -5 to +4).
  Richmond Agitation-Sedation Scale(scoring -5 to +4) is a valid and reliable instrument to assess level of sedation and agitated behavior during sedation.
level of sedation | 30 minutes after Ketamine injection
  assessed by Richmond Agitation-Sedation Scale(scoring -5 to +4).
  Richmond Agitation-Sedation Scale(scoring -5 to +4) is a valid and reliable instrument to assess level of sedation and agitated behavior during sedation.

SECONDARY OUTCOMES:
clinician's satisfaction | starts at the time of Ketamine injection through recovery period(maximum of 2 hours)
  assessed by a Clinician Satisfaction with Sedation Instrument(CSSI) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Sina Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sener S, Eken C, Schultz CH, Serinken M, Ozsarac M. Ketamine with and without midazolam for emergency department sedation in adults: a randomized controlled trial. Ann Emerg Med. 2011 Feb;57(2):109-114.e2. doi: 10.1016/j.annemergmed.2010.09.010. PMID 20970888
- [Background] Newton A, Fitton L. Intravenous ketamine for adult procedural sedation in the emergency department: a prospective cohort study. Emerg Med J. 2008 Aug;25(8):498-501. doi: 10.1136/emj.2007.053421. PMID 18660398
- [Background] Amr MA, Shams T, Al-Wadani H. Does haloperidol prophylaxis reduce ketamine-induced emergence delirium in children? Sultan Qaboos Univ Med J. 2013 May;13(2):256-62. doi: 10.12816/0003231. Epub 2013 May 9. PMID 23862031
- [Background] Chudnofsky CR, Weber JE, Stoyanoff PJ, Colone PD, Wilkerson MD, Hallinen DL, Jaggi FM, Boczar ME, Perry MA. A combination of midazolam and ketamine for procedural sedation and analgesia in adult emergency department patients. Acad Emerg Med. 2000 Mar;7(3):228-35. doi: 10.1111/j.1553-2712.2000.tb01064.x. PMID 10730829
- [Derived] Akhlaghi N, Payandemehr P, Yaseri M, Akhlaghi AA, Abdolrazaghnejad A. Premedication With Midazolam or Haloperidol to Prevent Recovery Agitation in Adults Undergoing Procedural Sedation With Ketamine: A Randomized Double-Blind Clinical Trial. Ann Emerg Med. 2019 May;73(5):462-469. doi: 10.1016/j.annemergmed.2018.11.016. Epub 2019 Jan 3. PMID 30611640